CLINICAL TRIAL: NCT06857799
Title: An Open-Label, Placebo-Controlled, Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Topical WS-0101 in Healthy Adult Subjects: a First-in-Human Clinical Trial
Brief Title: A Study on the Safety, Tolerability and Pharmacokinetics of WS-0101 Tablets in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Cui Yimin, Director of the Institute of Clinical Pharmacology, Director of the Clinical Trial Center, and Director of the Department of Pharmacy, Peking University, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS_WS-0101_101
Record Dates: First submitted 2024-10-11; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-05

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5% WS-0101/Placebo (Active Comparator): Treat with 5% WS-0101 medication or placebo.
  Interventions: Procedure: Light Power Density and Light Duration 40 mW/cm²*1000s; Procedure: Light Power Density and Light Duration 80 mW/cm²*1000s
- 10% WS-0101/Placebo (Active Comparator): Treat with 10% WS-0101 medication or placebo.
  Interventions: Procedure: Light Power Density and Light Duration 40 mW/cm²*1000s; Procedure: Light Power Density and Light Duration 80 mW/cm²*1000s
- 20% WS-0101/Placebo (Active Comparator): Treat with 20% WS-0101 medication or placebo.
  Interventions: Procedure: Light Power Density and Light Duration 80 mW/cm²*1000s

INTERVENTIONS:
Procedure: Light Power Density and Light Duration 40 mW/cm²*1000s — Use light power density and light duration 40 mW/cm²*1000s treatment
  Arms: 10% WS-0101/Placebo; 5% WS-0101/Placebo
Procedure: Light Power Density and Light Duration 80 mW/cm²*1000s — Use light power density and light duration 80 mW/cm²*1000s treatment

SUMMARY:
This study is an open-label, placebo-controlled, first-in-human clinical trial in healthy adults, designed to assess the safety, tolerability, and PK characteristics of various doses of WS-0101 following different light power density exposures. Each subject will receive the drug on the left upper arm and placebo on the right upper arm, followed by photodynamic therapy (PDT). Based on non-clinical results and considering systemic safety, the drug concentrations tested will be 5%, 10%, and 20%, and light power densities will be 40 and 80 mW/cm². The PDT equipment, provided by the sponsor, is the WS-L-01 device, with data on any related device defects collected for safety evaluation.

DETAILED DESCRIPTION:
Overall Study Design:

* Open-label, placebo-controlled, single-dose, dose-escalation study.
* The study includes 5 groups with varying drug concentrations and light power densities.

Group Drug Concentration Application Area Light Duration Light Power Density Sample Size 1-1 5% 3 cm diameter 1000 s 40 mW/cm² 3 1-2 5% 3 cm diameter 1000 s 80 mW/cm² 6 2-1 10% 3 cm diameter 1000 s 40 mW/cm² 6 2-2 10% 3 cm diameter 1000 s 80 mW/cm² 6 3 20% 3 cm diameter 1000 s 80 mW/cm² 6 Placebo Control: Self-controlled. Total Number of Subjects: 27 Dose Escalation Principles

1. The study will start with the lowest dose group, following the sequence shown in the table. If only one exploratory condition is added between groups, multiple dose groups may escalate simultaneously (e.g., Group 1-1 to Groups 1-2 and 2-1). After completing the observation of Group 2-1, the dose can escalate to Group 2-2, and after observing Group 2-2, it can proceed to Group 3.
2. Each dose group will be observed for at least 7 days following the first subject's dosing before escalating to the next group. The Safety Review Committee (SRC) will evaluate safety and tolerability before allowing progression to the next group.
3. The decision to move to the next dose level will be made by the SRC through a consensus decision-making process, which may involve meetings, teleconferences, or email responses. Specific processes will be detailed in a separate SRC charter.
4. Dose adjustments, either increases or decreases, will be based on the safety and tolerability results of the current group.

Possible adjustments to the planned dose escalation include:

* Lower than the starting dose.
* Intermediate doses between the current and preceding dose.
* Intermediate doses between the current and next planned dose.
* Repeat the current dose.
* Terminate further dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be included in this study:

  1. Voluntarily participate in the study and provide a signed and dated informed consent form (ICF).
  2. Be a male or female adult between 18 and 55 years of age (inclusive).
  3. Male subjects must weigh at least 50 kg, and female subjects must weigh at least 45 kg, with a body mass index (BMI) between 18.5 and 28 kg/m² (inclusive).
  4. For female subjects:

     1. No reproductive potential, including at least 6 weeks post-surgical sterilization (documented tubal ligation, hysterectomy, or bilateral oophorectomy) or ≥12 months of postmenopausal status (with follicle-stimulating hormone (FSH) levels ≥40 IU/L).
     2. For women of childbearing potential, they must be non-pregnant, non-lactating, and must agree to use non-drug contraceptive methods for 30 days before administration, throughout the study, and for 3 months after dosing. Their human chorionic gonadotropin (hCG) test must be negative at screening and on Day -1, and they must not donate eggs during this period.
  5. For male subjects with female partners of childbearing potential, they must agree to use non-drug contraceptive methods for 14 days before administration, throughout the study, and for 3 months after dosing. Male subjects must not donate sperm during this period.
  6. Willingness to comply with the study protocol, including visits, study treatment, laboratory tests, and other study-related procedures and requirements.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Known allergy to the study drug or its excipients, or allergy to blue light sources, or a history of severe allergies (including any food or drug allergies).
  2. A history of photosensitivity disorders, such as polymorphic light eruption, solar urticaria, chronic actinic dermatitis, porphyria, or any suspected photosensitivity based on the investigator's judgment.
  3. A history of recurrent skin infections, psychiatric disorders, a family history of psychiatric disorders, or chronic or serious conditions involving the central nervous system, cardiovascular system, liver, kidneys, lungs, digestive tract, metabolism, blood, or skeletal systems that could affect study participation or pose unacceptable risks.
  4. Sensitivity, infection, inflammation, redness, rash, sunburn, blistering, injury, pigmentation changes, or the presence of tattoos, birthmarks, or scars at the application site.
  5. Exposure of the upper arms to sunlight or artificial tanning within 48 hours prior to dosing.
  6. Keloid formation or scarring tendencies.
  7. Clinically significant abnormalities in vital signs, physical examination, or laboratory tests.
  8. Clinically significant abnormalities on a 12-lead electrocardiogram (ECG).
  9. A creatinine clearance rate (Ccr) of less than 90 mL/min, calculated using the Cockcroft-Gault formula: Ccr=((140-Age)*Weight(Kg)*(0.85 for women))/(72*Serum creatinine (mg/dL))

     Alternatively: Ccr=((140-Age)*Weight(Kg)*(0.85 for women))/(0.81*Serum creatinine (μmol/dL))
  10. Positive for human immunodeficiency virus antibodies (HIV-Ab), hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCV-Ab), or syphilis antibodies (TP-Ab).
  11. Use of any prescription, over-the-counter medication, herbal medicine, or dietary supplements within 14 days before dosing, or use of photosensitizing or phototoxic drugs (e.g., quinolones, glibenclamide, sulfonamides, tetracyclines, chloramphenicol, phenothiazines) within 3 months before dosing.
  12. Known or suspected history of substance abuse (e.g., morphine, methamphetamine, ketamine, MDMA, THC, cocaine), or a positive drug screen.
  13. Excessive alcohol consumption (more than 21 units per week; one unit equals 14 g alcohol, e.g., 360 mL of 5% beer, 45 mL of 40% spirits, or 120 mL of 12% wine) within 1 year prior to screening, or a positive alcohol breath test.
  14. Smoking more than 5 cigarettes per day within 3 months prior to screening, or an inability to comply with the study's smoking restrictions.
  15. Daily consumption of more than 6 servings of caffeine (e.g., coffee, tea, cola, energy drinks) within 3 months prior to screening, or consumption of caffeine-containing products within 24 hours prior to dosing.
  16. Participation in another clinical trial within the past 3 months.
  17. Recent or planned surgery within the study period.
  18. Receipt of a vaccine within 30 days prior to screening, or a planned vaccine during the study.
  19. Blood donation or significant blood loss (≥400 mL) within 1 month prior to screening, or planned blood donation during the study.
  20. Inability to tolerate venipuncture for blood collection, or a history of fainting or phobias related to blood draws.
  21. Unwillingness to assist with photographic documentation of the application site.
  22. Any other condition or circumstance deemed by the investigator to make participation in the study inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of different topical doses of WS-0101, followed by varying light power densities, in healthy adult subjects | Visit 11 (Day14)
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0, Change From Baseline in Pain Scores on the Numerical Rating Scale (NRS) at 2 Weeks

SECONDARY OUTCOMES:
Assess PK characteristics of single-dose topical WS-0101 in healthy adults and evaluate the safety of the laser therapy device based on defect incidence | Visit 6 (Day 1)
  Non-compartmental analysis using WinNonlin will be used to estimate PK parameters such as Cmax, AUC0-t, AUC0-∞, and Tmax. Descriptive statistics for Cmax, AUC0-t, Tmax, and other parameters will be provided and listed. Boxplots will be drawn for key PK parameters such as Cmax, AUC0-t, and AUC0-∞ by dose group. If plasma exposure is too low and there are insufficient quantifiable concentrations to calculate relevant PK parameters, only concentration data and/or partial parameters will be listed.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.trialos.com.cn